CLINICAL TRIAL: NCT06796374
Title: A Comparison of Fisetin Kinetics in Young and Old Adults - FISEKIN-1
Brief Title: A Comparison of Fisetin Kinetics in Young and Old Adults
Acronym: FISEKIN-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IPHA-2025-010
Record Dates: First submitted 2025-01-13; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Pharmacokinetic Study in Healthy Volunteers
MeSH Terms: interventions — fisetin; Quercetin

STUDY DESIGN:
Intervention Model Description: The kinetic study will be designed as an open-label, two-cohorts (young vs. old), four-arm, randomized cross-over, single oral dose protocol.
Masking Description: This study is an opel-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 2: Fisetin - Cohort 2: old age (≥ 65 years) (Active Comparator)
  Interventions: Dietary Supplement: Fisetin
- Arm 4: Fisetin + Quercetin - Cohort 2: old age (≥ 65 years) (Active Comparator)
  Interventions: Dietary Supplement: Fisetin + Quercetin
- Arm 1: Fisetin - Cohort 1: young age (18-30 years) (Active Comparator)
  Interventions: Dietary Supplement: Fisetin
- Arm 3: Fisetin + Quercetin - Cohort 1: young age (18-30 years) (Active Comparator)
  Interventions: Dietary Supplement: Fisetin + Quercetin

INTERVENTIONS:
Dietary Supplement: Fisetin — A single oral dose of 100 mg fisetin (as Novusetin®) will be administered as 1 capsule with 240 ml of still water in the overnight fasting condition:
  A total of 18 blood samples will be taken at defined time points (baseline; 10; 20; 30; 40; 50; 60; 80; 100 min; 2.0; 2.5; 3.0; 4.0; 5.0; 6.0; 8.0; 10.0; 24.0 h). At each time point, blood will be collected (4.9 ml for separation of plasma) to determine fisetin, and fisetin metabolites. The total amount of blood collected for each participant and each arm is 90 ml at the kinetic visits and 12 ml at the screening visit. Urine will be collected during the first 10 hours after fisetin administration.
  Arms: Arm 1: Fisetin - Cohort 1: young age (18-30 years); Arm 2: Fisetin - Cohort 2: old age (≥ 65 years)
Dietary Supplement: Fisetin + Quercetin — A single oral dose of 1000 mg fisetin + 200 mg quercetin will be administered as 2 softgel capsule with 240 ml of still water in the overnight fasting condition:
  A total of 18 blood samples will be taken at defined time points (baseline; 10; 20; 30; 40; 50; 60; 80; 100 min; 2.0; 2.5; 3.0; 4.0; 5.0; 6.0; 8.0; 10.0; 24.0 h). At each time point, blood will be collected (4.9 ml for separation of plasma) to determine fisetin, fisetin metabolites, and quercetin. The total amount of blood collected for each participant and each arm is 90 ml at the kinetic visits and 12 ml at the screening visit. Urine will be collected during the first 10 hours after fisetin administration.
  Arms: Arm 3: Fisetin + Quercetin - Cohort 1: young age (18-30 years); Arm 4: Fisetin + Quercetin - Cohort 2: old age (≥ 65 years)

SUMMARY:
This study investigates the differences in the kinetic parameters of fisetin in two cohorts of healthy volunteers:

Cohort 1) volunteers aged 18-30 years (n = 40) Cohort 2) volunteers aged 65 years or older (n = 40)

The purpose of this study is:

1. To describe the fisetin kinetics after a single dose oral administration in older age.
2. To compare the fisetin kinetics after a single dose oral administration in old and young age.

FISEKIN-1 is designed as a four-arm study protocol. As well as two different age groups (18-30 years vs. 65 years and older), we want to compare fisetin kinetic parameters in two different fisetin formulations and dosages :

Arm 1) 100 mg fisetin (1x 1 capsule), cohort 1: young age Arm 2) 100 mg fisetin (1x 1 capsule), cohort 2: old age Arm 3) 1000 mg fisetin + 200 mg quercetin (2x 1 softgel capsule), cohort 1: young age Arm 4) 1000 mg fisetin + 200 mg quercetin (2x 1 softgel capsule), cohort 2: old age

DETAILED DESCRIPTION:
The study is designed as an open-label, two-cohorts (young vs. old), four-arm, cross-over, single oral dose protocol.

A single oral dose of fisetin will be administered as capsules with 240 ml of still water in the overnight fasting condition.

Both arms will be conducted in each participant in random order with a wash-out period of at least one week between each arm.

A total of 18 blood samples will be taken at defined time points (baseline; 10; 20; 30; 40; 50; 60; 80; 100 min; 2.0; 2.5; 3.0; 4.0; 5.0; 6.0; 8.0; 10.0; 24.0 h). At each time point, blood will be collected (4.9 ml for separation of plasma) to determine fisetin, its metabolites, and quercetin (only in arm 3 and 4).

The total amount of blood collected for each participant and each arm is 90 ml at the kinetic visits and 12 ml at the screening visit.

After intake of fisetin, participants will drink 200 ml of sparkling water every hour to stimulate gastrointestinal peristalsis and to promote transport of the capsule. After 2 hours, the participants may drink a cup of tea or coffee and after 4 hours they will be served a meal low in fisetin content. Urine will be collected during the first 10 hours after fisetin administration. Monitoring of blood pressure and heart rate will take place for the first 4 hours after administration. Volunteers will stay in the Clinical Research Unit of the Institute of Pharmacology for the first 10 hours after administration.

ELIGIBILITY:
Inclusion Criteria:

* any sex
* age between 18 and 30 years or ≥ 65 years
* understands the study purpose and design
* contractually capable and provides signed informed consent form
* healthy condition or mild and/or well-treated forms of allergies, asthma, hypertension, and orthopedic diseases
* a maximum of 3 chronically taken drugs

Exclusion Criteria:

* BMI > 30 kg/m2 and < 18 kg/m2
* body weight < 48 kg
* women in young cohort: known pregnancy or lactation period; positive urine pregnancy test at screening or kinetic visit
* men: hemoglobin < 13 g/dl (8,07 mmol/l) women: hemoglobin < 12 g/dl (7,45 mmol/l)
* elevated liver function tests (1 or more of ALAT, ASAT, yGT, Bilirubin > 2x ULN)
* reduced renal function (eGFRMDRD < 60 ml/min/1,7 m2)
* QTcF > 450 ms in screening ECG
* psychiatric disease requiring recent or actual treatment
* drug dependency at the time of visit
* use of recreational drugs more than twice a week
* any known hypersensitivity or allergic reactions to fisetin
* history of severe hypersensitivity reactions and/or anaphylaxis
* poor venous conditions that make it impossible to place a peripheral venous catheter and regularly draw blood through it
* intake of drugs interfering with CYP1A2, CYP2D6, CYP2C8, CYP2C9, CYP2C19, CYP3A4, and/or Pgp during the past seven days if the duration of intake was at least two days
* individuals who have eaten food with high fisetin content in the two days before the kinetic visits (e.g. strawberry, apple, persimmon, grape, mango, kiwi, peach, tomato, onion, lotus roots, kale, cucumber; processed products, e.g. wine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Fisetin plasma concentration arm 1 vs. arm 2 | 24 hours
  Difference of fisetin plasma concentrations between the young and old cohort, expressed as area under the curve (AUC0-24h).
Fisetin plasma concentration arm 3 vs. arm 4 | 24 hours
  Difference of fisetin plasma concentrations between the young and old cohort, expressed as area under the curve (AUC0-24h).

SECONDARY OUTCOMES:
Fisetin metabolites plasma concentration arm 1 vs. arm 2 | 24 hours
  Difference in plasma concentrations of fisetin metabolites between the young and old cohort, expressed as area under the curve (AUC0-24h).
Fisetin metabolites plasma concentration arm 3 vs. arm 4 | 24 hours
  Difference in plasma concentrations of fisetin metabolites between the young and old cohort, expressed as area under the curve (AUC0-24h).
Fisetin plasma concentration arm 1 vs. arm 2 | 24 hours
  Difference plasma concentrations of fisetin and fisetin metabolites between the young and old cohort, expressed as maximum plasma concentration (Cmax).
Fisetin plasma concentration arm 3 vs. arm 4 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between the young and old cohort, expressed as maximum plasma concentration (Cmax).
Fisetin plasma concentration arm 1 vs. arm 2 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between the young and old cohort, expressed as time at maximum concentration (Tmax).
Fisetin plasma concentration arm 3 vs. arm 4 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between the young and old cohort, expressed as time at maximum concentration (Tmax).
Fisetin plasma concentration arm 1 vs. arm 2 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between the young and old cohort, expressed as total clearance.
Fisetin plasma concentration arm 3 vs. arm 4 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between the young and old cohort, expressed as total clearance.
Fisetin plasma concentration arm 1 vs. arm 2 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between the young and old cohort, expressed as renal clearance.
Fisetin plasma concentration arm 3 vs. arm 4 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between the young and old cohort, expressed as renal clearance.
Fisetin plasma concentration arm 1 vs. arm 2 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between the young and old cohort, expressed as apparent volume of distribution.
Fisetin plasma concentration arm 3 vs. arm 4 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between the young and old cohort, expressed as apparent volume of distribution.
Fisetin plasma concentration arm 1 vs. arm 3 | 24 hours
  Difference of fisetin plasma concentrations between arm 1 and arm 3, expressed as area under the curve (AUC0-24h).
Fisetin plasma concentration arm 2 vs. arm 4 | 24 hours
  Difference of fisetin plasma concentrations between arm 2 and arm 4, expressed as area under the curve (AUC0-24h).
Fisetin plasma concentration arm 1 vs. arm 3 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between arm 1 and arm 3, expressed as maximum plasma concentration (Cmax).
Fisetin plasma concentration arm 2 vs. arm 4 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between arm 2 and arm 4, expressed as maximum plasma concentration (Cmax).
Fisetin plasma concentration arm 1 vs. arm 3 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between arm 1 and arm 3, expressed as time at maximum concentration (Tmax).
Fisetin plasma concentration arm 2 vs. arm 4 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between arm 2 and arm 4, expressed as time at maximum concentration (Tmax).
Fisetin plasma concentration arm 1 vs. arm 3 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between arm 1 and arm 3, expressed as total clearance.
Fisetin plasma concentration arm 2 vs. arm 4 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between arm 2 and arm 4, expressed as total clearance.
Fisetin plasma concentration arm 1 vs. arm 3 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between arm 1 and arm 3, expressed as renal clearance.
Fisetin plasma concentration arm 2 vs. arm 4 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between arm 2 and arm 4, expressed as renal clearance.
Fisetin plasma concentration arm 1 vs. arm 3 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between arm 1 and arm 3, expressed as apparent volume of distribution.
Fisetin plasma concentration arm 2 vs. arm 4 | 24 hours
  Difference in plasma concentrations of fisetin and fisetin metabolites between arm 2 and arm 4, expressed as apparent volume of distribution.
Quercetin plasma concentration arm 3 vs. arm 4 | 24 hours
  Difference of quercetin plasma concentrations between the young and old cohort, expressed as area under the curve (AUC0-24h).
Quercetin plasma concentration arm 3 vs. arm 4 | 24 hours
  Difference of quercetin plasma concentrations between the young and old cohort, expressed as maximum plasma concentration (Cmax).
Quercetin plasma concentration arm 3 vs. arm 4 | 24 hours
  Difference of quercetin plasma concentrations between the young and old cohort, expressed as time at maximum concentration (Tmax).
Quercetin plasma concentration arm 3 vs. arm 4 | 24 hours
  Difference of quercetin plasma concentrations between the young and old cohort, expressed as total clearance.
Quercetin plasma concentration arm 3 vs. arm 4 | 24 hours
  Difference of quercetin plasma concentrations between the young and old cohort, expressed as renal clearance.
Quercetin plasma concentration arm 3 vs. arm 4 | 24 hours
  Difference of quercetin plasma concentrations between the young and old cohort, expressed as apparent volume of distribution.

IPD SHARING:
Plan to Share IPD: No